CLINICAL TRIAL: NCT03016910
Title: Coronary Artery Plaque Burden in Type 2 Diabetes Mellitus. Changes Over Time, Relation to Risk Profile, and Comparison to Acute Myocardial Infarction.
Brief Title: Coronary Artery Plaque Burden and Morphology in Type 2 Diabetes Mellitus.
Acronym: CARPEDIEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Svendborg Hospital (Other)
Responsible Party: Principal Investigator, Laurits Heinsen, Medical doctor, Svendborg Hospital
Other Study IDs: CD20150029
Record Dates: First submitted 2017-01-02; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Type2 Diabetes; Atherosclerosis; Plaque, Atherosclerotic; Plaque Vulnerability; Diabetes Complications; Microalbuminuria; Coronary Computed Tomography Angiography
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic; Diabetes Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be stored at -80 degrees celcius for a biobank. These includes:
  5 x 2 ml (serum).
  4 x 2 ml (ethylenediaminetetraacetic acid "EDTA").
  2 x 2 ml (sodium citrate)
  1 x 2 ml (buffy coat)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 2 diabetes: This group will consist of 300 patients with type 2 diabetes mellitus without symptoms or known coronary heart disease. The group will be followed for one year and CCTA will be performed at baseline and after one year.
- Type 1 diabetes: This group will consist of 50-100 patients with type 1 diabetes mellitus without symptoms or known coronary heart disease. The group will be followed for one year. CCTA will be performed at baseline and after one year.

SUMMARY:
Unstable plaque, the primary cause of myocardial infarction, is characterized by distinct a morphology including positive remodeling (PR), low attenuated plaque (LAP), napkin ring sign (NRS), and spotty calcifications (SC) The purpose of the present study is to investigate the influence of microvascular dysfunction and additional risk factors on plaque morphology and plaque burden in patients with diabetes mellitus.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death and morbidity in type 2 diabetes mellitus (T2DM) and diabetics holds the same risk for death or myocardial infarction (MI) as patients with a prior (MI) without diabetes. In addition to macrovascular complications, and traditional cardiac risk factors, T2DM is burdened by microvascular dysfunction affecting several organs. The dynamics between microvascular dysfunction, known cardiac risk factors and coronary atherosclerosis in diabetic disease is not well characterized.

In the present study, a primary cohort of 300 type 2 diabetics and a subgroup of 50-100 type 1 diabetics will be examined with CCTA at baseline and after one year. In addition, CAD in diabetes will be compared to a historical cohort of patients with acute myocardial infarction (AMI).

All study participant will undergo the following examinations at baseline:

* CCTA
* CAC-score
* Transthoracic echocardiography
* 12-lead ECG
* Blood pressure and pulse frequency
* Height, weight, waist to hip-ratio
* Blood samples and urin samples
* Medical history

After 12 months all of the above examinations will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Type 1 or 2 diabetes mellitus
* Ability to provide informed conscent

Exclusion Criteria:

* History of CAD
* Symtoms of CAD (angina)
* Any tachyarrhythmias making CCTA impossible
* Glumerular filtration rate (GFR)< 45 ml/min
* Allergy to iodine contrast
* Critical illness with life expectancy less than 1 year
* Documented heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 1 or 2 diabetes mellitus without history of CAD or relevant symptoms (angina). Patients are recruited at the out-patient clinic at Svendborg Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Changes in plaque burden stratified by diabetic complications. | Baseline,12 months.
  Changes in plaque burden (percentage) during 12 months in diabetics with or without diabetic complications.
Changes in plaque burden stratified by cardiovascular risk factors | Baseline, 12 months
  Changes in plaque burden during 12 months stratified by cardiovascular risk factors (hypertension,hypercholersterolemia, smoking, overweight/obesity)
Changes in plaque morphology stratified by diabetic complications | Baseline, 12 months
  Changes in plaque morphology (PR, LAP, NRS, SC) during 12 months in diabetics either with or without diabetic complications.
Changes in plaque morphology stratified by cardiovascular risk factors. | Baseline,12 months
  Changes in plaque burden during 12-months stratified by cardiovascular risk factors

SECONDARY OUTCOMES:
Changes in plaque burden in diabetes compared to AMI-patients without diabetes. | Baseline and 12 months
  A comparison of plaque burden (percentage) in diabetes and a historical cohort of AMI-patients.
Changes in plaque morphology in diabetes compared to AMI-patients without diabetes. | Baseline,12-months
  A comparison of plaque morphology in diabetes and a historical cohort of AMI-patients.
Changes in plaque burden during 12 months in relation to HbA1c and cholesterol levels. | Baseline,12-months
  Changes in plaque burden during 12 months stratified by historical levels of cholesterol and HbA1c levels recorded from onset of diabetes to present.
Changes in plaque morphology during 12 months in relation to HbA1c and cholesterol levels. | Baseline,12-months
  Changes in plaque morphology during 12 months stratified by historical levels of cholesterol and HbA1c levels recorded once a year from onset of diabetes to present.
Impact of asymtomatic CAD in diabetes on future events. | 5-7 years
  Long term follow-up to evaluate the impact of asymptomatic CAD (plaque burden and morphology) in diabetes on death, coronary heart attack, hospitalization due to unstable angina, heart failure and ischemic stroke.
  Clinical outcomes will be recorded from journal records and analyzed after 5-7 years.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, Prof. DMSci, Study Director — Head of Reseach, Cardiovascular Research Unit, OUH Svendborg Hospital
Locations (1):
- University Hospital of Odense (OUH) Svendborg Hospital, Svendborg, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinsen LJ, Pararajasingam G, Andersen TR, Auscher S, Sheta HM, Precht H, Lambrechtsen J, Egstrup K. High-risk coronary artery plaque in asymptomatic patients with type 2 diabetes: clinical risk factors and coronary artery calcium score. Cardiovasc Diabetol. 2021 Aug 9;20(1):164. doi: 10.1186/s12933-021-01350-2. PMID 34372839